CLINICAL TRIAL: NCT01509482
Title: Insulin Resistance : a New Diagnosis of the Pathogenesis of Idiopathic Oligozoospermia and Non Obstructive Azoospermia
Brief Title: Insulin Resistance in Idiopathic Oligospermia and Azoospermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Egyptian IVF-ET Center (Other)
Responsible Party: Principal Investigator, Ragaa Mansour, Director, the Egyptian IVF-ET center, The Egyptian IVF-ET Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: insulin resistance
Record Dates: First submitted 2012-01-06; First posted 2012-01-13 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Insulin Resistance; Oligospermia; Azoospermia
Keywords: insulin resistance; unexplained azoospermia; unexplained oligospermia
MeSH Terms: conditions — Insulin Resistance; Oligospermia; Azoospermia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- insulin resistance (Experimental): unexplained oligospermia and azoospermia. Blood samples will be taken for hormonal and blood lipids analysis.
  Interventions: Other: blood samples
- Fertile males (Active Comparator): Healthy Men with proven fertility. Blood samples will be taken for hormonal and blood lipids analysis
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: blood samples — blood samples to test for primary and secondary outcome measures
  Other Names: Unexplained oligospermia and azoospermia
  Arms: insulin resistance
Other: Blood samples — IR Cholesterol HDL LDL Fasting Glucose Triglycerides
  Other Names: Hypospermatogenesis
  Arms: Fertile males

SUMMARY:
Insulin resistance in men can be the underlying major factor in reproductive abnormalities ( chronic hypospermatogenesis ) as well as metabolic abnormalities similar to polycystic ovarian syndrome ( PCOS ) in women.

DETAILED DESCRIPTION:
During the past decade IR has been recognized as a major contributor to the pathogenesis of chronic anovulation, hyperandrogenism and metabolic abnormalities associated with PCOS . Theoretically IR in men may result in a similar reproductive abnormalities ( chronic hypospermatogenesis ) as well as other metabolic abnormalities similar to what happens in PCOS in women .

ELIGIBILITY:
Inclusion Criteria:

* sperm count less than 10 million per milliliter
* non-obstructive azoospermia

Exclusion Criteria:

* high FSH ( > 10 mIU/ ml )
* high prolactin ( > 36 mIU/ml )
* abnormal karyotype
* AZF

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
serum insulin | one month

SECONDARY OUTCOMES:
Fasting Glucose | one month
cholesterol | one month
high density lipoprotein ( HDL) | one month
Low density lipoprotein ( LDL ) | one month
testosterone | one month
Triglycerides | One month

CONTACTS AND LOCATIONS:
Overall Officials: Ragaa Mansour, MD,PhD, Principal Investigator — The Egyptian IVF-ET Center
Locations (1):
- The Egyptian IVF-ET center, Cairo, Egypt, Egypt